CLINICAL TRIAL: NCT03254043
Title: Evaluating a Novel Medication Device for Methadone Dosing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00145200; R34DA042926-01A1 (NIH)
Record Dates: First submitted 2017-08-09; First posted 2017-08-18 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment-as-Usual (Active Comparator): Participants will routine methadone clinic care.
  Interventions: Behavioral: Take-home Dosing Procedures
- Take-home Dosing using MedMinder "Jon" Electronic Pill Box (Experimental): Participants will receive 50% of their methadone dose in the morning in the clinic and 50% of their dose will be dispensed in an electronic pill box for participants to take at home later that day.
  Interventions: Behavioral: Take-home Dosing Procedures
- Choice Phase (Other): Participants will be allowed to select one final Treatment-As-Usual or the MedMinder "Jon" Electronic Pill Box for the final phase of the study.
  Interventions: Behavioral: Take-home Dosing Procedures

INTERVENTIONS:
Behavioral: Take-home Dosing Procedures — Within-subject evaluation across 2 phases with a final choice condition

SUMMARY:
This study will evaluate whether a commercially available, secure, electronic pill box is a feasible, acceptable, and satisfactory method to manage take-home dosing of methadone for both methadone clinic patients and staff members.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Receiving methadone for the treatment of opioid use disorder for at least 90 days and having been on the same methadone dose for at least 30 days
* Have previously received a take-home dose of methadone as part of routine care
* Be willing to comply with the study schedule
* Be a methadone patient in the clinic within which this study is being conducted

Exclusion Criteria:

* Pregnancy
* Presence of an acute medical problems that requires immediate or intense medical management
* Presence of serious or unstable mental illness that interferes with study procedures
* Planning to leave methadone treatment within the next 12 weeks
* Being maintained on a dose of methadone that is less than 10mg or more than 100mg
* Currently receiving split doses of methadone as part of routine care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Participant willingness to use the MedMinder "Jon" electronic pillbox to manage take-home doses of methadone | Week 12
  Feasibility will be assessed by conducting a survival analysis of participant retention in the study
Participant acceptance of the MedMinder "Jon" electronic pillbox to manage take-home doses of methadone | Week 9
  Percent of participants who select the Electronic Pill Box during their Choice phase (phase 3)
Change in participant satisfaction | Week 4
  Participant satisfaction will be assessed using the Client Satisfaction Questionnaire- an 8-item self-report measure on which patients will rate their satisfaction with treatment on a 4-item Likert scale. Values will be summed for a total satisfaction rating (range 8-32), with higher scores indicating greater satisfaction. Participants will complete the CSQ at week 4 and week 8, and the CSQ ratings from the treatment-as-usual will be subtracted from the ratings following the MedMinder "Jon" electronic pillbox phase as a measure of change in participant satisfaction.
Change in participant satisfaction | Week 8
  Participant satisfaction will be assessed using the Client Satisfaction Questionnaire- an 8-item self-report measure on which patients will rate their satisfaction with treatment on a 4-item Likert scale. Values will be summed for a total satisfaction rating (range 8-32), with higher scores indicating greater satisfaction. Participants will complete the CSQ at week 4 and week 8, and the CSQ ratings from the treatment-as-usual will be subtracted from the ratings following the MedMinder "Jon" electronic pillbox phase as a measure of change in participant satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dunn, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services (ATS), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No